CLINICAL TRIAL: NCT06272994
Title: Swab Testing to Optimize Pneumonia Treatment with Empiric Vancomycin (STOP-Vanc)
Brief Title: Swab Testing to Optimize Pneumonia Treatment with Empiric Vancomycin
Acronym: STOP-Vanc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey A Freiberg, Assistant Professor of Medicine, Division of Infectious Diseases, MD, PhD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231724
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Community-acquired Pneumonia
Keywords: MRSA; Vancomycin; Nasal Swab
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: This study will be performed as a single center, pragmatic, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No MRSA Nasal Swab (No Intervention): Subjects will not have a nasal swab collected.
- MRSA Nasal Swab (Active Comparator): Subjects will have a nasal swab collected and sent to the clinical laboratory for the MRSA nasal swab PCR test to be run. For the subjects assigned to the intervention group who have a negative MRSA nasal swab PCR result, providers will receive a pager alert which inform them of the negative result and will direct clinicians to clinical guidance recommending clinicians to discontinue vancomycin, if clinically appropriate.
  Interventions: Diagnostic Test: MRSA Nasal Swab PCR

INTERVENTIONS:
Diagnostic Test: MRSA Nasal Swab PCR — For the subjects assigned to the intervention group who have a negative MRSA nasal swab PCR result, providers will receive a pager alert which inform them of the negative result and will direct clinicians to clinical guidance recommending clinicians to discontinue vancomycin, if clinically appropriate.
  Arms: MRSA Nasal Swab

SUMMARY:
This is a single center, pragmatic, randomized clinical trial (pRCT) examining whether reporting the results of a negative rapid PCR back to the provider via a pager alert results in decreased vancomycin utilization for critically ill adults with community-acquired pneumonia when compared with usual care.

DETAILED DESCRIPTION:
Methicillin-resistant Staphylococcus aureus (MRSA) is a critical antimicrobial resistant threat responsible for greater than 300,000 inpatient infections and 15,000 deaths per year in the United States. Community-acquired pneumonia (CAP) is a major driver of hospital antibiotic use. Nationally, there are around 600,000 CAP-related hospital admissions annually. However, MRSA is an infrequent cause of community-acquired pneumonia (CAP), accounting for less than 1% of cases. Despite this, MRSA is a frequently feared cause of CAP, which leads to the frequent use of vancomycin, an anti-MRSA antibiotic, in empiric CAP treatment.

Inappropriate antibiotic use can lead to avoidable adverse drug events and costs, as well as drive antimicrobial resistance. Empiric vancomycin use in patients hospitalized for pneumonia has demonstrated increased mortality, acute kidney injury (AKI), and secondary infections. The use of vancomycin is unfortunately associated with a high risk for toxicity and serious adverse events. Up to two-thirds of patients receiving high dose vancomycin develop AKI. Additionally, bone marrow suppression, linear IgA bullous dermatosis, anaphylaxis, and life-threatening hypersensitivity reactions are seen with vancomycin use. Furthermore, vancomycin is a costly antibiotic to use in the hospital as it requires careful monitoring due to its narrow therapeutic range and high risk of toxicity.

There is growing data to support the use of MRSA nasal swabs as a screening method to guide de-escalation of vancomycin use in CAP. A 2018 meta-analysis found using nasal swabs for MRSA screening had an overall 96.5% negative predictive value (NPV) for pneumonia, which was increased to 98.1% among patients with CAP or Healthcare-associated pneumonia (HCAP). Multiple retrospective studies along with one prospective study utilizing MRSA nasal swab-based de-escalation protocols have shown MRSA nasal swab use to be effective in decreasing vancomycin use and associated costs without having any negative effects on patient outcomes. Among these studies, significant decreases in hospital length of stay and rate of AKI have been shown. Furthermore, the use of MRSA detection in nasal swabs is now consistent with guideline-based management of CAP. However, all the aforementioned studies are quasi-experimental analyses. To date there are no randomized controlled studies of the use of MRSA nasal swab guided antibiotic de-escalation.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age greater than or equal to 18) patients admitted/transferred to the Vanderbilt University Medical Center (VUMC) Medical Intensive Care Unit (MICU) from the VUMC Emergency Department or from a hospital floor within 48 hours of admission.
* Suspicion for pneumonia on admission (defined as an indication for antibiotics of "respiratory infection" and/or an order for a respiratory culture i.e., sputum culture, tracheal aspirate culture, or bronchoalveolar lavage (BAL) culture).
* No topical nasal decolonization during hospitalization prior to collection of MRSA nasal swab PCR.
* Must match both of the following in either order:

  * The patient has been admitted to and physically located in the MICU.
  * The patient has received a continuing vancomycin order, or a pharmacokinetics consult for a continuing vancomycin order, no later than 24 hours following their physical admission to the MICU.

Exclusion Criteria:

* Hospital stay of longer than 48 hours prior to MICU admission.
* Known to be a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Vancomycin-free hours alive | Baseline to seven days following enrollment.
  The number of hours out of the seven days following enrollment in the trial that the patient is alive and not receiving vancomycin estimated using a proportional odds ratio model with the ordinal status levels being alive and not on vancomycin, alive and on vancomycin, or dead.

SECONDARY OUTCOMES:
Time Alive off Vancomycin | Baseline to seven days following enrollment.
  The number of hours out of the 168 hours (7 days) following enrollment in the trial that the patient is alive and not receiving vancomycin.
30-day all-cause mortality | Thirty days following enrollment.
  Mortality within 30 days with date of study enrollment as day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Freiberg, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Jernigan JA, Hatfield KM, Wolford H, Nelson RE, Olubajo B, Reddy SC, McCarthy N, Paul P, McDonald LC, Kallen A, Fiore A, Craig M, Baggs J. Multidrug-Resistant Bacterial Infections in U.S. Hospitalized Patients, 2012-2017. N Engl J Med. 2020 Apr 2;382(14):1309-1319. doi: 10.1056/NEJMoa1914433. PMID 32242356
- [Background] Klein EY, Jiang W, Mojica N, Tseng KK, McNeill R, Cosgrove SE, Perl TM. National Costs Associated With Methicillin-Susceptible and Methicillin-Resistant Staphylococcus aureus Hospitalizations in the United States, 2010-2014. Clin Infect Dis. 2019 Jan 1;68(1):22-28. doi: 10.1093/cid/ciy399. PMID 29762662
- [Background] Jones BE, Ying J, Stevens V, Haroldsen C, He T, Nevers M, Christensen MA, Nelson RE, Stoddard GJ, Sauer BC, Yarbrough PM, Jones MM, Goetz MB, Greene T, Samore MH. Empirical Anti-MRSA vs Standard Antibiotic Therapy and Risk of 30-Day Mortality in Patients Hospitalized for Pneumonia. JAMA Intern Med. 2020 Apr 1;180(4):552-560. doi: 10.1001/jamainternmed.2019.7495. PMID 32065604
- [Background] Tongsai S, Koomanachai P. The safety and efficacy of high versus low vancomycin trough levels in the treatment of patients with infections caused by methicillin-resistant Staphylococcus aureus: a meta-analysis. BMC Res Notes. 2016 Sep 29;9(1):455. doi: 10.1186/s13104-016-2252-7. PMID 27686168
- [Background] van Hal SJ, Paterson DL, Lodise TP. Systematic review and meta-analysis of vancomycin-induced nephrotoxicity associated with dosing schedules that maintain troughs between 15 and 20 milligrams per liter. Antimicrob Agents Chemother. 2013 Feb;57(2):734-44. doi: 10.1128/AAC.01568-12. Epub 2012 Nov 19. PMID 23165462
- [Background] Fortuna G, Salas-Alanis JC, Guidetti E, Marinkovich MP. A critical reappraisal of the current data on drug-induced linear immunoglobulin A bullous dermatosis: a real and separate nosological entity? J Am Acad Dermatol. 2012 Jun;66(6):988-94. doi: 10.1016/j.jaad.2011.09.018. Epub 2011 Dec 9. PMID 22169257
- [Background] Madigan LM, Fox LP. Vancomycin-associated drug-induced hypersensitivity syndrome. J Am Acad Dermatol. 2019 Jul;81(1):123-128. doi: 10.1016/j.jaad.2019.02.002. Epub 2019 Feb 6. PMID 30738120
- [Background] Huang V, Clayton NA, Welker KH. Glycopeptide Hypersensitivity and Adverse Reactions. Pharmacy (Basel). 2020 Apr 21;8(2):70. doi: 10.3390/pharmacy8020070. PMID 32326261
- [Background] Wilhelm MP. Vancomycin. Mayo Clin Proc. 1991 Nov;66(11):1165-70. doi: 10.1016/s0025-6196(12)65799-1. PMID 1943250
- [Background] Rybak MJ, Le J, Lodise TP, Levine DP, Bradley JS, Liu C, Mueller BA, Pai MP, Wong-Beringer A, Rotschafer JC, Rodvold KA, Maples HD, Lomaestro BM. Therapeutic monitoring of vancomycin for serious methicillin-resistant Staphylococcus aureus infections: A revised consensus guideline and review by the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, the Pediatric Infectious Diseases Society, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2020 May 19;77(11):835-864. doi: 10.1093/ajhp/zxaa036. No abstract available. PMID 32191793
- [Background] Parente DM, Cunha CB, Mylonakis E, Timbrook TT. The Clinical Utility of Methicillin-Resistant Staphylococcus aureus (MRSA) Nasal Screening to Rule Out MRSA Pneumonia: A Diagnostic Meta-analysis With Antimicrobial Stewardship Implications. Clin Infect Dis. 2018 Jun 18;67(1):1-7. doi: 10.1093/cid/ciy024. PMID 29340593
- [Background] Dadzie P, Dietrich T, Ashurst J. Impact of a Pharmacist-driven Methicillin-resistant Staphylococcus aureus Polymerase Chain Reaction Nasal Swab Protocol on the De-escalation of Empiric Vancomycin in Patients with Pneumonia in a Rural Healthcare Setting. Cureus. 2019 Dec 13;11(12):e6378. doi: 10.7759/cureus.6378. PMID 31938656
- [Background] Huffman V, Andrade DC, Ham J, Brown K, Melnitsky L, Lopez Cohen A, Parmar J. Impact of Nasal Swabs on Empiric Treatment of Respiratory Tract Infections (INSERT-RTI). Pharmacy (Basel). 2020 Jun 11;8(2):101. doi: 10.3390/pharmacy8020101. PMID 32545231
- [Background] Woolever NL, Schomberg RJ, Cai S, Dierkhising RA, Dababneh AS, Kujak RC. Pharmacist-Driven MRSA Nasal PCR Screening and the Duration of Empirical Vancomycin Therapy for Suspected MRSA Respiratory Tract Infections. Mayo Clin Proc Innov Qual Outcomes. 2020 Aug 15;4(5):550-556. doi: 10.1016/j.mayocpiqo.2020.05.002. eCollection 2020 Oct. PMID 33083704
- [Background] Dunaway S, Orwig KW, Arbogast ZQ, Myers ZL, Sizemore JA, Giancola SE. Evaluation of a pharmacy-driven methicillin-resistant Staphylococcus aureus surveillance protocol in pneumonia. Int J Clin Pharm. 2018 Jun;40(3):526-532. doi: 10.1007/s11096-018-0647-3. Epub 2018 May 2. PMID 29721739
- [Background] Smith MN, Erdman MJ, Ferreira JA, Aldridge P, Jankowski CA. Clinical utility of methicillin-resistant Staphylococcus aureus nasal polymerase chain reaction assay in critically ill patients with nosocomial pneumonia. J Crit Care. 2017 Apr;38:168-171. doi: 10.1016/j.jcrc.2016.11.008. Epub 2016 Nov 15. PMID 27918901
- [Background] Willis C, Allen B, Tucker C, Rottman K, Epps K. Impact of a pharmacist-driven methicillin-resistant Staphylococcus aureus surveillance protocol. Am J Health Syst Pharm. 2017 Nov 1;74(21):1765-1773. doi: 10.2146/ajhp160964. PMID 29070498
- [Background] Baby N, Faust AC, Smith T, Sheperd LA, Knoll L, Goodman EL. Nasal Methicillin-Resistant Staphylococcus aureus (MRSA) PCR Testing Reduces the Duration of MRSA-Targeted Therapy in Patients with Suspected MRSA Pneumonia. Antimicrob Agents Chemother. 2017 Mar 24;61(4):e02432-16. doi: 10.1128/AAC.02432-16. Print 2017 Apr. PMID 28137813
- [Background] Diep C, Meng L, Pourali S, Hitchcock MM, Alegria W, Swayngim R, Ran R, Banaei N, Deresinski S, Holubar M. Effect of rapid methicillin-resistant Staphylococcus aureus nasal polymerase chain reaction screening on vancomycin use in the intensive care unit. Am J Health Syst Pharm. 2021 Dec 9;78(24):2236-2244. doi: 10.1093/ajhp/zxab296. PMID 34297040
- [Background] Raush N, Betthauser KD, Shen K, Krekel T, Kollef MH. Prospective Nasal Screening for Methicillin-Resistant Staphylococcus aureus in Critically Ill Patients With Suspected Pneumonia. Open Forum Infect Dis. 2021 Nov 19;9(1):ofab578. doi: 10.1093/ofid/ofab578. eCollection 2022 Jan. PMID 34988251
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Self WH, Wunderink RG, Williams DJ, Zhu Y, Anderson EJ, Balk RA, Fakhran SS, Chappell JD, Casimir G, Courtney DM, Trabue C, Waterer GW, Bramley A, Magill S, Jain S, Edwards KM, Grijalva CG. Staphylococcus aureus Community-acquired Pneumonia: Prevalence, Clinical Characteristics, and Outcomes. Clin Infect Dis. 2016 Aug 1;63(3):300-9. doi: 10.1093/cid/ciw300. Epub 2016 May 8. PMID 27161775
- [Derived] Freiberg JA, Siemann JK, Qian ET, Ereshefsky BJ, Hennessy C, Stollings JL, Rali TM, Harrell FE, Gatto CL, Rice TW, Nelson GE; Vanderbilt Center for Learning Healthcare. Swab Testing to Optimize Pneumonia treatment with empiric Vancomycin (STOP-Vanc): study protocol for a randomized controlled trial. Trials. 2024 Dec 28;25(1):854. doi: 10.1186/s13063-024-08705-6. PMID 39732716
- [Derived] Freiberg JA, Siemann JK, Qian ET, Ereshefsky BJ, Hennessy C, Stollings JL, Rali TM, Harrell FE, Gatto CL, Rice TW, Nelson GE; Vanderbilt Center for Learning Healthcare. Swab Testing to Optimize Pneumonia treatment with empiric Vancomycin (STOP-Vanc): study protocol for a randomized controlled trial. Res Sq [Preprint]. 2024 Jun 18:rs.3.rs-4365928. doi: 10.21203/rs.3.rs-4365928/v1. PMID 38947088